CLINICAL TRIAL: NCT06433687
Title: HeakHeart Phase 1 Proof of Concept Study
Brief Title: Evaluation of the HekaHeart Platform in Medication Management for Heart Failure Patients
Acronym: HekaHeart POC
Status: Withdrawn | Type: Observational
Why Stopped: Not funded.
Sponsor: Yale University (Other)
Collaborators: HekaHeart (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000037817
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Guideline-directed medical therapy; Remote monitoring; Medication optimization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HekaHeart-based medication optimization and remote monitoring: Patients will onboard to the HekaHeart platform, which will recommend a GDMT management plan that has been validated by a Yale-based clinician, with consideration given to eligibility for GDMT, past medical history, and patient preference. Participants will also be provided with an at-home blood pressure cuff, weight scale, and heart rate monitor and be instructed to use these devices on a regular cadence. Measurements will be electronically transmitted in real-time to the HekaHeart platform and uploaded to a web-based portal for review. Weekly/bi-weekly scheduled remote check-ins will be used by clinicians to monitor patient progress with GDMT management, to evaluate whether additional medications or dose adjustments are necessary, monitor symptoms, identify issues, offer medical education, and provide continued assistance with remote patient monitoring (RPM) devices. A final patient offboarding visit will occur once the patient has been on the platform for 45 days.
  Interventions: Device: HekaHeart platform medication management and remote monitoring

INTERVENTIONS:
Device: HekaHeart platform medication management and remote monitoring — Onboarding to the HekaHeart platform which includes a personalized GDMT management plan along with remote monitoring kits including a scale, blood pressure cuff, and heart rate monitor. Patients engage in video and phone calls with clinicians who will use established standardized clinical protocols to guide medication and vital optimization. Once patients are determined to be maximally titrated on all GDMT, they are transitioned back to standard clinical care.

SUMMARY:
This pilot study will test the feasibility of a novel digital health technology-enabled platform, HekaHeart, developed to facilitate comprehensive medical management, including medication initiation, titration, e-prescription eligibility, remote patient monitoring, and communication of care coordination activities, for patients with Heart Failure with Reduced Ejection Fraction (HFrEF) not currently on all four pillars of guideline-directed medical therapy (GDMT).

DETAILED DESCRIPTION:
Heart Failure (HF) is a major cause of morbidity, mortality, and healthcare expenditure in the United States (US). The 2022 AHA/ACC/HFSA Guideline for the management of HF strongly recommends quadruple therapy for all patients with HFrEF, which includes: beta-blockers (BB); renin-angiotensin-aldosterone-system (RAAS) inhibitors such as angiotensin-converting enzyme inhibitors (ACEi), angiotensin receptor blockers (ARB) and angiotensin receptor-neprilysin inhibitors (ARNi); mineralocorticoid receptor antagonists (MRA); and sodium-glucose cotransporter-2 inhibitors (SGLT2i). Unfortunately, suboptimal adoption of GDMT persists despite mounting, unambiguous evidence of its substantial benefit on patient outcomes (including mortality) across numerous large-scale studies.

Further, following initial prescription of quadruple therapy, augmentation of each pillar to target or highest tolerated dosing is critical to achieve maximum benefit, as shown in a recent multinational randomized controlled trial (STRONG-HF) where rapid uptitration to optimal doses of GDMT reduced the risk of death and hospitalization just 180 days after an acute HF episode. Yet, multiple contemporary registry studies continue to reflect suboptimal uptake and dose escalation of GDMT for patients with HFrEF in real-world clinical practice due to both clinical and patient-based barriers.

The HekaHeart platform is a comprehensive remote care and monitoring-based method for GDMT titration and management. The platform uses a virtual team of clinicians with expertise in HF to manage GDMT prescription, dose escalation, and symptom monitoring for patients with HFrEF as a means to both provide personalized patient care and support while alleviating clinician burden. Once a patient is fully optimized with respect to GDMT, they are transitioned back to routine clinical care.

The present study will evaluate the usability of the HekaHeart platform to initiate, monitor, and manage GDMT for patients with HFrEF. The study will prospectively recruit eligible patients from ambulatory HF clinics affiliated with Yale New Haven Health System (YNHHS). Consented patients will be onboarded to the HekaHeart platform for GDMT management by HF disease management clinicians, which will include medication adjustment and remote patient monitoring to assess laboratory results, changes in body weight, blood pressure, and heart rate. Throughout the study, patients will engage in short message service (SMS), video and phone check-ins with clinicians, who will leverage standardized titration protocols to guide medication optimization, monitor patient progress and symptoms, and collect, analyze and respond to remote monitoring data. After 45 days, patients will be transitioned back to usual care.

The primary outcome is the Net Promoter Score (NPS), collected at study offboarding by each participant, and used to assess patient satisfaction with the HekaHeart platform and experience. The secondary outcome is the increase in proportion of HFrEF patients prescribed four pillars of GDMT. Other secondary endpoints include percent of patients successfully onboarded to the HekaHeart platform, proportion of patients whose GDMT is titrated toward target or maximally tolerated dosing, number scheduled visits attended, and percent of platform GDMT recommendations implemented.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HFrEF as evidenced by the presence of LVEF ≤40% reading at any time within the last 12 months,

  1. with associated symptoms of HF
  2. or an elevated NT-proBNP
  3. or a hospitalization for HF within the preceding 12 months
* Currently receiving care at YNHHS
* Currently not on all 4 recommended classes of GDMT (BB, ACEi/ARB/ARNi, MRA, and SGLT2i)

Exclusion Criteria:

* Currently pregnant or breast feeding
* Received or listed for cardiac transplantation
* Planned or present durable left ventricular-assist device (LVAD)
* Goals of treatment are palliation
* Currently has a condition(s) that limit survival to <1 year
* Unable to provide informed consent
* Unwilling to use remote monitoring devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will come from two outpatient Heart Failure clinics associated with Yale New Haven Hospital. The population will be adults ≥18 years with symptomatic HFrEF who are not on adequate GDMT.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Net Promoter Score | Assessed at time off patient offboarding (45 days after enrollment)
  A metric used to gauge patient satisfaction with the HekaHeart platform. Patients are asked how likely they are to recommend the platform to a friend on a scale of 1 to 10 (with 1 being not likely to recommend, and 10 being highly likely to recommend).

SECONDARY OUTCOMES:
Percent of patients on all eligible guideline-directed medical therapy (GDMT) classes | Assessed at time off patient offboarding (45 days after enrollment)
  Patients assessed for number of eligible classes of eligible GDMT medications prescribed.
Percent of enrolled patients onboarded to HekaHeart | Assessed from time of enrollment to 45 days post-enrollment
  Percent of patients who consented to the study who have successfully onboarded to the HekaHeart plan with an optimized medication management plan.
Percent of onboarded patients successfully prescribed a new medication | Assessed from time of enrollment to 45 days post-enrollment
  Percent of patients who have been prescribed a new medication within the HekaHeart platform after enrollment.
Percent of scheduled study check-ins attended by patients | Assessed from time of enrollment to 45 days post-enrollment
  Percent of patients who attended a scheduled check-in (via SMS, text, email, or phone)
Percent of medication recommendations implemented | Assessed from time of enrollment to 45 days post-enrollment
  Percent of HekaHeart-recommended medications prescribed
Time to maximum titration | Assessed from time of enrollment to 45 days post-enrollment
  Time in days to optimal titration of all eligible classes of GDMT as determined by clinician judgement and expertise
Time from patient enrollment to first remote prescription | Assessed from time of enrollment to 45 days post-enrollment
  Time in days to first prescription made in HekaHeart platform
Ease of implementation of HekaHeart platform | Assessed up to one month post- study completion
  Determined via qualitative survey assessment of clinicians which asks how well the HekaHeart platform integrates into existing systems and workflows

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Shoreline Medical Center- 111 Goose Lane location, Guilford, Connecticut
  - Yale Physicians Building- 800 Howard Ave location, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for the primary and secondary outcomes will be made available upon publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available upon publication and indefinitely.